CLINICAL TRIAL: NCT00580775
Title: Effects of Early Hormone Replacement Therapy on Risk Factors for Sudden Cardiac Death: Autonomic Function and Ventricular Repolarization Heterogeneity ( A KEEPS Ancillary Study)
Brief Title: Study of Early Hormone Replacement Therapy on Risk Factors for Sudden Cardiac Death
Acronym: KEEPS
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Rachel Lampert, Associate Professor of Medicine, Yale University
Other Study IDs: 0505000069
Record Dates: First submitted 2007-12-19; First posted 2007-12-27 (Estimated); Last update posted 2015-01-22 (Estimated); Status verified 2015-01

CONDITIONS: Menopausal Women
Keywords: Menopause; Hormone Replacement Therapy; Sudden Cardiac Death
MeSH Terms: conditions — Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Placebo: Observing heart rate variability in placebo and active estrogen preparations
- Active estogen: Observing heart rate variability in placebo and active estrogen preparations

SUMMARY:
As an ancillary study to the KEEPS study (see ClinicalTrials.gov Identifier: NCT00154180), the primary purpose is to measure effects of estrogen vs. placebo in menopausal women, on autonomic function and repolarization; both measured non-invasively via holter monitoring.

DETAILED DESCRIPTION:
The parent study KEEPS, will be a randomized, placebo-controlled double blinded, prospective trial with two active groups and one placebo group. Only patients enrolled in KEEPS will be invited to participate in this ancillary study.Duration of the KEEPS study will be for 4 years after randomization for each study subject, with assessment of the primary endpoint, carotid CIMT, twice at baseline, 12, 24, 36 and 48 months. Ancillary to the KEEPS study, patients will undergo holter monitoring at baseline, 24 and 48 months.Data will be analyzed after 24 and 48 months (corresponding to data analysis of the primary endpoints.) Holter monitors will be put on during the scheduled KEEPS visits, will be worn for 24 hours and will be returned the following day. Effects of estrogen on heart rate variability (HRV) and repolarization parameters will be evaluated, and also correlated with clinical, quality of life, sleep and mood information gathered through the parent study. Anticipated enrollment from the parent study at this site is 90 study subjects. This ancillary does not involve the use of drugs or investigational devices.

ELIGIBILITY:
Inclusion Criteria:

* participant of the KEEPS parent study: ClinicalTrials.gov Identifier NCT00154180

Exclusion Criteria:

* non-participants of parent study

Ages: 42 Years to 58 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Self-voluntary study subjects participating in the KEEPS parent study which is randomized, double-blind, placebo controlled.
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2005-09; Primary Completion 2008-07 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Heart rate variability | 48 Months

SECONDARY OUTCOMES:
Repolarization parameters | 48 Months

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Lampert, M.D., Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine / Yale New Haven Hospital, New Haven, Connecticut, United States